CLINICAL TRIAL: NCT01751074
Title: A Two-Part, Open-label, Sequential, Double Cohort, Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Rosuvastatin When Co Administered With Darapladib in Healthy Adult Subjects
Brief Title: To Estimate the Potential Effects of Repeat Doses of Darapladib on the Pharmacokinetics (PK) of Rosuvastatin as Well as Evaluating Safety and Tolerability in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115677
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Atherosclerosis
Keywords: Drug interaction, rosuvastatin, healthy volunteer, Lp-PLA2, atherosclerosis, darapladib, pharmacokinetics.
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium; darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): All subjects will be of Caucasian descent and will receive single dose of Rosuvastatin 10 mg for 1 day (Day 1) during treatment period 1, then will receive Darapladib 160 mg once daily (QD) for 10 days (Day 5 to 14) in treatment period 2. Immediately following this, all subjects will receive the combination of Darapladib 160 mg and Rosuvastatin 10 mg for 1 day (Day 15) and continued Darapladib dosing of 160 mg QD for additional 3 days (Days 16 to 18) in treatment period 2.
  Interventions: Drug: Rosuvastatin 10 mg; Drug: Darapladib 160 mg
- Part B (Experimental): The decision to initiate Part B will be made by the GSK study team based on an evaluation of data from Part A. Part B will consist of a cohort of healthy subjects of Far-East Asian descent and will be conducted similar to Part A.
  Interventions: Drug: Rosuvastatin 10 mg; Drug: Darapladib 160 mg

INTERVENTIONS:
Drug: Rosuvastatin 10 mg — Enteric coated tablet will be administered orally as a single dose once in Treatment Period 1 (Day 1) and Treatment Period 2 (Day 15).
  Other Names: Crestor
Drug: Darapladib 160 mg — Enteric coated tablet will be administered orally as once daily for 14 days in Treatment Period 2 only (Day 5 to Day 18).

SUMMARY:
The potential for a drug interaction between Darapladib and Rosuvastatin is felt to be low and it would be helpful to quantify this risk in man in order to guide prescribing physicians. The primary aims of this study are to estimate the potential effects of repeat doses of Darapladib on the PK of Rosuvastatin as well as evaluating safety and tolerability. Two part approaches are planned for this study. Part A of the study will examine the effects of repeat doses Darapladib on the PK of Rosuvastatin in healthy volunteers of Caucasian descent. Based on whether a significant increase in Rosuvastatin exposure is observed in Caucasians in Part A, a decision will be made regarding whether to proceed with a conditional Part B to examine this effect in healthy volunteers of Far-East Asian descent.

In both parts, subjects will receive Rosuvastatin 10 milligrams (mg) once daily (QD) for 1 day during the first treatment period (Treatment Period 1), followed by a 4 day PK sampling period/wash-out. Subjects will then receive darapladib 160 mg QD for the next 10 days with 24-hour PK sampling on the last day (Day 14 of the study). Immediately following this, all subjects will then receive the combination of Darapladib 160 mg and Rosuvastatin 10 mg for 1 day and continued Darapladib dosing of 160 mg QD for additional 3 days (Treatment Period 2) while blood samples are collected to assess Rosuvastatin PK. Plasma samples collected on Day 15 will be analyzed for both Rosuvastatin and Darapladib concentrations.

Subjects will be required to return to the unit approximately 10 to 14 days following the last dose of study medication for a clinic visit for assessments and then will return again at 35 ±7 days following the last dose for the final follow-up visit of the study. The duration of each subject's participation in the study from screening to follow-up will be approximately three months.

Approximately 18 evaluable subjects will be enrolled in Part A and another 18 subjects will be enrolled in Part B (if conducted) to complete dosing and all assessments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 20 and 64 years of age inclusive, at the time of signing the informed consent.
* Subject must be of Caucasian or of Far-East Asian Descent. Far -East Asian is defined as a person of self-reported Asian ancestry including that of Japanese, Korean or Chinese descent (which includes Taiwanese subjects) [for Part B only].
* Far East Asian subjects must have been born in their native countries and have resided less than 10 years outside their native countries [for Part B only].
* Far East Asian subjects must have maintained a lifestyle, including diet, without significant change since leaving his/her native country [for Part B only].
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone > 40 milliliter of urine (MlU)/ milliliter (mL) and estradiol < 40 picogram/mL (<147 picomoles/liter is confirmatory] or Child-bearing potential and is abstinent or agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until follow-up.
* Body mass index within the range 19 to 37 kilogram/meter^2 (inclusive)

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* A positive pre-study drug/alcohol screen.
* A positive test for human immune virus (HIV) antibody
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: Thirty days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in a previous study or donor bank would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Requiring the use of oral or injectable strong cytochrom P3A4 inhibitors.
* Pregnant females as determined by positive human chorionic gonadotropin test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or history of heparin-induced thrombocytopenia.
* History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions Clinical criteria for diagnosing anaphylaxis or severe allergic responses.
* Consumption of grapefruit or grapefruit juice >8 ounce within 7 days prior to the first dose of study medication

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2013-03-14 (Actual); Study Completion 2013-03-14 (Actual)

PRIMARY OUTCOMES:
Single dose PK of Rosuvastatin assessed by AUC (0-infinity) or AUC (0-t) when co-administered with darapladib and when administered alone. | 09 days. Blood samples will be collected on Day 1 to 5 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 hours [hrs] post dose) and on Day 15 to 18 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 24, 36, 48, 72, and 96 hrs post dose).
  To evaluate the single dose PK of Rosuvastatin, area under the concentration-time curve from time zero extrapolated to infinite time (AUC [0-infinity]) or area under the concentration-time curve from time zero to last time of quantifiable concentration (AUC [0-t]) will be assessed.
Single dose PK of Rosuvastatin assessed by Cmax when co-administered with darapladib and when administered alone. | 09 days. Blood samples will be collected on Day 1 to 5 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 hours [hrs] post dose) and on Day 15 to 18 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 24, 36, 48, 72, and 96 hrs post dose).
  To evaluate the single dose PK of Rosuvastatin, maximum observed concentration (Cmax) will be assessed.
Single dose PK of Rosuvastatin assessed by Tmax and T1/2 (as data permit) when co-administered with darapladib and when administered alone. | 09 days. Blood samples will be collected on Day 1 to 5 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 hours [hrs] post dose) and on Day 15 to 18 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 24, 36, 48, 72, and 96 hrs post dose).
  To evaluate the single dose PK of Rosuvastatin, time of occurrence of Cmax (Tmax), and terminal phase half-life (T1/2) will be assessed.

SECONDARY OUTCOMES:
Single dose Rosuvastatin PK compared between Caucasian subjects (Part A) and if performed, Asian subjects (Part B). | 05 days. Blood samples will be collected on Day 1 to Day 5 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours [hrs] post dose).
  Single dose Rosuvastatin PK will be assessed by comparison of AUC (0-infinity), or AUC (0-t), Cmax, Tmax and T1/2 as data permit.
Rosuvastatin PK when co-administered with repeat doses of Darapladib compared between Caucasian subjects (Part A) and if performed, Asian subjects (Part B). | 01 day. Blood samples will be collected on Day 15 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hrs post dose) of each part.
  Rosuvastatin PK when co-administered with repeat doses of Darapladib will be assessed by comparison of AUC (0-infinity), or AUC (0-t), Cmax, Tmax and T1/2 as data permit.
Repeat doses PK of Darapladib compared between Caucasian subjects (Part A) and if performed, Asian subjects (Part B). | 02 days. Blood samples will be collected on Day 13 (pre-dose), and Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hrs post-dose) of each part.
  Repeat doses PK of Darapladib assessed by comparison of area under the concentration-time curve over the dosing interval (AUC [0-tau]), Cmax, Tmax and T1/2 as data permit
Repeat doses PK of Darapladib assessed by AUC (0-tau) when co-administered with single dose of Rosuvastatin and when administered alone. | 03 days. Blood samples will be collected on Day 13 (pre-dose), Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hrs post-dose) and Day 15 (0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hrs post dose).
  To evaluate the repeat doses PK of Darapladib, AUC (0-tau), will be assessed when repeat doses of Darapladib given with single dose of Rosuvastatin and when given alone.
Repeat doses PK of Darapladib assessed by Cmax when co-administered with single dose Rosuvastatin and when administered alone | 03 days. Blood samples will be collected on Day 13 (pre-dose), Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hrs post-dose) and Day 15 (0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hrs post dose).
  To evaluate the repeat doses PK of Darapladib, Cmax will be assessed when repeat doses of Darapladib given with single dose of Rosuvastatin and when given alone.
Repeat doses PK of Darapladib assessed by Tmax, and T1/2 (as data permit) when co-administered with Rosuvastatin and when administered alone | 03 days. Blood samples will be collected on Day 13 (pre-dose), Day 14 (pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12 and 24 hrs post-dose) and Day 15 (0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hrs post dose).
  To evaluate the repeat doses PK of Darapladib, Tmax, and T1/2 will be assessed when repeat doses of Darapladib given with single dose of Rosuvastatin and when given alone.
Safety and tolerability of darapladib when co-administered with Rosuvastatin assessed by incidence and severity of adverse events | Up to 60 days
  Adverse events (AEs) will be collected from the start of study treatment and until the follow-up contact. Intensity of AEs will be categorized as mild, moderate or severe
Safety and tolerability of darapladib when co-administered with Rosuvastatin assessed by vital signs | Up to 60 days
  Vital signs measurement will include systolic and diastolic blood pressure and pulse rate.
Safety and tolerability of darapladib when co-administered with Rosuvastatin assessed by clinical laboratory data | Up to 60 days
  Clinical laboratory tests include hematology, clinical chemistry, urinalysis and additional parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115677 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115677?search=study&search_terms=115677#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register